CLINICAL TRIAL: NCT03852680
Title: Current Treatment Modalities for Wide Necked Intracranial Aneurysms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdalla Ragab Abdelrahman Morsy, Assisstant lecturer of neurosurgery, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Intracranial aneurysms
Record Dates: First submitted 2019-02-10; First posted 2019-02-25 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Brain Aneurysm
Keywords: wide necked intracranial aneurysms
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: aneurysm clipping — treatment of wide necked intracranial aneurysms using different modalities as open surgery by clipping or endovascular techniques as coiling and flow diversion
  Other Names: aneurysm coiling; flow diversion

SUMMARY:
* Give an effective treatment for intracranial wide necked aneurysm and can detect the best method could be used.
* Improve the outcome of these patients and decease rate of recurrence and complications.

DETAILED DESCRIPTION:
The prevalence of intracranial aneurysms in the adult population is estimated to be around 2 %. Most remain asymptomatic, but there is a risk of rupture of 1.2 % per year, and this risk increases in line with the diameter of the aneurysm. If rupture occurs, subarachnoid hemorrhage and its associated acute complications are responsible for high mortality (between 30 and 67 %) and morbidity (between 15 and 30 %).

Coil embolization of intracranial aneurysms has made remarkable technological progress since the International Subarachnoid Aneurysm Trial (ISAT) data were released in 2005. However, wide-necked aneurysms remain a great challenge to be treated via the endovascular means, as they are associated with a significantly greater incidence of adverse events when compared with narrow-necked ones.

Acutely ruptured wide-necked intracranial aneurysms pose technical challenges to the treating physician; thus, multiple endovascular techniques have been described to treat these lesions, including balloon-assisted coil placement, double microcatheter technique, and microcatheter assisted coil placement. However, the use of these techniques can sometimes be limited, owing to the lack of permanent support for the coil mass inside the aneurysm sac, which may lead to coil prolapse or migration after the procedure, especially for wide-necked aneurysms (dome-to-neck ratio is less than 1) or tiny aneurysms (3 mm). Therefore, surgical clipping is preferred for acutely ruptured wide-necked intracranial aneurysms in most institutions. Surgery, however, may also be challenging in some of these lesions, since clips may slip, and surgical access may be limited because of the swelling of the brain in the acute setting of a subarachnoid hemorrhage.

Flow diverters are new implantable medical devices that make possible to embolize wide-necked aneurysms without the use of coils; the efficacy results published to date are encouraging in terms of complete occlusion in the medium-term, thereby confirming the innovative nature of the flow diversion technique that we aim to evaluate without the use of coils.

ELIGIBILITY:
Inclusion Criteria:

• Patients who undergo surgical clipping or any endovascular techniques used in treatment of wide-necked intracranial aneurysms. Wide-necked aneurysms are defined as aneurysms with a fundus-to-neck ratio of less than 2 or a neck diameter of 14 mm.

Exclusion Criteria:

* patients with narrow-necked intracranial aneurysms
* patients who are unfit for any neurosurgical interventions.
* patients who had artery aneurysm and vascular malformation due to some trauma.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-08-01 (Estimated); Study Completion 2021-03-30 (Estimated)

PRIMARY OUTCOMES:
Independent clinical outcome changes | one day before treatment, within 3 days after treatment.
  The changes in clinical condition of the patients will be assessed before and after treatment using modified Rankin scale, as the scale runs from 0-6, running from perfect health without symptoms to death.
  0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead.
Postoperative angiographic occlusion rate changes | within 3 days after treatment and after 6 months
  The changes in postoperative angiographic occlusion rate will be assessed in different time frame using CT angiography or conventional angiography (if CT angiography is not conclusive)

SECONDARY OUTCOMES:
incidence of aneurysm rupture | during operation or within 7 days after treatment
  as complication of treatment
incidence of cerebral vasospasm | within 30 days after treatment
  as complication of treatment
Mortality rate | within 30 days after treatment
  as a result of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Ahmed Abokresha, Assisstant professor, Study Director — Assiut University; Mohamed El-Sayed Mahmoud, Assisstant professor, Study Director — Assiut University; Abd El-hai Moussa Abd El-Latif, professor of neurosurgery, Study Chair — Assiut University
Locations (1):
- Faculty of medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brown RD Jr, Broderick JP. Unruptured intracranial aneurysms: epidemiology, natural history, management options, and familial screening. Lancet Neurol. 2014 Apr;13(4):393-404. doi: 10.1016/S1474-4422(14)70015-8. PMID 24646873
- [Background] Wermer MJ, van der Schaaf IC, Algra A, Rinkel GJ. Risk of rupture of unruptured intracranial aneurysms in relation to patient and aneurysm characteristics: an updated meta-analysis. Stroke. 2007 Apr;38(4):1404-10. doi: 10.1161/01.STR.0000260955.51401.cd. Epub 2007 Mar 1. PMID 17332442
- [Background] Matillon Y. [Ruptured intracranial aneurysms: Occlusion by endovascular approach versus exclusion by microsurgery]. J Radiol. 2002 May;83(5):662-4. No abstract available. French. PMID 12063434
- [Background] Layton KF, Cloft HJ, Gray LA, Lewis DA, Kallmes DF. Balloon-assisted coiling of intracranial aneurysms: evaluation of local thrombus formation and symptomatic thromboembolic complications. AJNR Am J Neuroradiol. 2007 Jun-Jul;28(6):1172-5. doi: 10.3174/ajnr.A0490. PMID 17569982
- [Background] Moret J, Cognard C, Weill A, Castaings L, Rey A. The "Remodelling Technique" in the Treatment of Wide Neck Intracranial Aneurysms. Angiographic Results and Clinical Follow-up in 56 Cases. Interv Neuroradiol. 1997 Mar 30;3(1):21-35. doi: 10.1177/159101999700300103. Epub 2001 May 15. PMID 20678369
- [Background] Baxter BW, Rosso D, Lownie SP. Double microcatheter technique for detachable coil treatment of large, wide-necked intracranial aneurysms. AJNR Am J Neuroradiol. 1998 Jun-Jul;19(6):1176-8. PMID 9672035
- [Background] Ihn YK, Kim DI, Kim BS, Lee JM. Utility of catheter-assisted Guglielmi detachable coiling in the treatment of wide-necked aneurysms. Acta Neurochir (Wien). 2006 Oct;148(10):1045-52; discussion 1052. doi: 10.1007/s00701-006-0881-7. Epub 2006 Sep 8. PMID 16944050
- [Background] Gory B, Sigovan M, Vallecilla C, Courbebaisse G, Turjman F. High-resolution MRI visualization of aneurysmal thrombosis after flow diverter stent placement. J Neuroimaging. 2015 Mar-Apr;25(2):310-311. doi: 10.1111/jon.12110. Epub 2014 Mar 19. PMID 24641489
- [Background] Brinjikji W, Murad MH, Lanzino G, Cloft HJ, Kallmes DF. Endovascular treatment of intracranial aneurysms with flow diverters: a meta-analysis. Stroke. 2013 Feb;44(2):442-7. doi: 10.1161/STROKEAHA.112.678151. Epub 2013 Jan 15. PMID 23321438